CLINICAL TRIAL: NCT00950092
Title: Numeris-AF Tethered Coagulation System With VisiTrax Indicated For Treatment of Persistent and Longstanding Persistent Atrial Fibrillation
Brief Title: nContactSurgical Numeris-AF Tethered Coagulation System for Treatment of Persistent & LSP AF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: nContact Surgical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VAL-1116(C)
Record Dates: First submitted 2009-07-29; First posted 2009-07-31 (Estimated); Last update posted 2014-04-03 (Estimated); Status verified 2013-09

CONDITIONS: Atrial Fibrillation
Keywords: AF; atrial fibrillation; ablation; surgical ablation; afib; coagulation; RF; epicardial; Arrhythmias
MeSH Terms: conditions — Atrial Fibrillation; Thrombosis; Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Other)
  Interventions: Device: Numeris-AF Tethered Coagulation System with VisiTrax

INTERVENTIONS:
Device: Numeris-AF Tethered Coagulation System with VisiTrax — Surgical radiofrequency (RF) epicardial ablation using the nContact Numeris-AF Tethered Coagulation System
  Other Names: RF Ablation; Coagulation of cardiac tissue; nContact Surgical

SUMMARY:
This is a multi center, non-randomized, prospective, open label, clinical trial evaluating the safety and efficacy of the nContact Surgical Numeris-AF Tethered Coagulation System when used to treat patients with persistent and longstanding persistent AF during concomitant cardiac surgery.

DETAILED DESCRIPTION:
The purpose of this study is to determine the safety and efficacy of the Numeris-AF Tethered Coagulation System with VisiTrax when used to treat persistent and longstanding persistent Atrial Fibrillation(AF)during concomitant cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years; < 80 years
* Left atrium =< 6.0 cm
* Documented persistent or longstanding persistent AF
* History of AF =< 10 years
* Scheduled for a concomitant cardiac procedure

  * Coronary bypass surgery (CABG)
  * Mitral valve repair/replacement
  * Aortic valve replacement
  * ASD repair
  * Tricuspid valve repair/replacement
  * Myxoma
  * Any combination of the above procedures
* Provided written informed consent

Exclusion Criteria:

* Left atrial size > 6.0 cm (pre-op TTE - parasternal 4 chamber view)
* History of AF > 10 years
* Left ventricular ejection fraction < 30%
* Pregnant or planning to become pregnant during study
* Co-morbid medical conditions that limit one year life expectancy
* History of coagulopathy
* Patients who are contraindicated for anticoagulants(heparin, warfarin etc.)
* Previous cardiac surgery
* History of pericarditis
* Previous cerebrovascular accident (CVA)
* Patients who have active infection or sepsis
* Patients who have uncorrected reversible cause(s) of AF such as hyperthyroidism and electrolyte imbalance
* Patients who are being treated for ventricular arrhythmias
* Patients who have had a previous catheter ablation for AF (does not include ablation for Aflutter)
* Current participation in another clinical investigation of a medical device or a drug, or recent participation in such a study within 30 days prior to study enrollment.
* Not competent to legally represent him or herself (e.g., requires a guardian or caretaker as a legal representative).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-10; Primary Completion 2013-06 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
The primary effectiveness endpoint will be assessed as number of subjects free from AF and free of all Class I and III Anti Arrhythmic Drugs (AADs) through 9 months post procedure. | 9 months

SECONDARY OUTCOMES:
Secondary effectiveness endpoint: Proportion of subjects free from AF regardless of their Class I and III AADs status through 9 months post procedure. | 9 months
Secondary effectiveness endpoint: Proportion of subjects free of AF/ AFL / AT and off all Class I and Class III AADs. | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Edward Garrett, M.D., Principal Investigator — Baptist Memorial Hospital - Memphis
Locations (2):
- United States (2):
  - Venice Regional Medical Center, Venice, Florida
  - Baptist Memorial Hospital, Memphis, Tennessee